CLINICAL TRIAL: NCT05331833
Title: Omitting Clinical Target Volume Under PET-CT Guidance in Unresectable Stage III Non-small-cell Lung Cancer.
Brief Title: Omitting Clinical Target Volume of Unresectable Stage III Non-small-cell Lung Cancer.
Status: Completed | Type: Observational
Sponsor: Jianguo Sun (Other)
Responsible Party: Sponsor-Investigator, Jianguo Sun, Clinical Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Other Study IDs: XQonc-018
Record Dates: First submitted 2022-03-29; First posted 2022-04-18 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Stage III Non-small-cell Lung Cancer
Keywords: PET-CT; IMRT; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: CTV-omitted IMRT under PET-CT guidance
  Interventions: Radiation: The enrollment was randomly (1:1) assigned into the study group with CTV-omitted IMRT under PET-CT guidance and the control group with CTV-delineated IMRT using a random number table.
- control group: CTV-delineated IMRT under PET-CT guidance
  Interventions: Radiation: The enrollment was randomly (1:1) assigned into the study group with CTV-omitted IMRT under PET-CT guidance and the control group with CTV-delineated IMRT using a random number table.

INTERVENTIONS:
Radiation: The enrollment was randomly (1:1) assigned into the study group with CTV-omitted IMRT under PET-CT guidance and the control group with CTV-delineated IMRT using a random number table.

SUMMARY:
About 20-30% of patients with stage III non-small cell lung cancer (NSCLC) are unresectable and definitive concurrent radiochemotherapy is the standard care. Intensity-modulated radiation therapy (IMRT) is a new radiotherapy technology, including gross tumor volume (GTV), clinical target volume (CTV), internal target volume (ITV), and planning target volume (PTV) as delineated target volumes. The treatment failure of local advanced NSCLC is mainly caused by local recurrence accounted for 50% and distant metastasis accounted for 50%. Local recurrence occurs both within the radiation field and outside the radiation field. Elective nodal irradiation (ENI) was designed before, however the adverse events (AEs) was not satisfactory. Afterwards, involved field radiotherapy (IFRT) showed that a reduced irradiation field did not increase local recurrence, and lowered the AEs Thus, IFRT has been broadly used in clinical work instead of ENI. IFRT still has disadvantages, including the risk of radiation respiratory events and radiation esophagitis, can the irradiation area be further reduced to reduce adverse reactions without affecting the efficacy? Positron emission tomography -computed tomography (PET-CT) can accurately assess primary tumor and metastatic lymph nodes in NSCLC patients better than CT . A meta-analysis of 39 clinical studies showed that the median sensitivity and specificity of PET-CT for the detection of lymph node involvement were 85% and 90%, respectively, while those of CT alone were only 61% and 79%, respectively. The radiotherapy application of PET-CT in image acquisition can ensure the delineation of both primary tumor and mediastinal lymph node metastasis. Under this condition, can the radiation field be further reduced to lower the dose to normal tissue and radiotherapy-associated AEs? A dosimetry study showed that when a dose of 60 Gy was given to the primary tumor and positive mediastinal lymph nodes, even if the CTV was omitted, a dose of 50 Gy was sufficient to cover the subclinical area.

DETAILED DESCRIPTION:
A dosimetry study showed that when a dose of 60 Gy was given to the primary tumor and positive mediastinal lymph nodes, even if the CTV was omitted, a dose of 50 Gy was sufficient to cover the subclinical area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced (Stage IIIA or IIIB AJCC 7) NSCLC that was histologically or cytologically inoperable
* ECOG whole body status (performancestatus,PS) level 0 or 1
* The estimated survival time is more than 12 weeks, 18 ~75 years old
* Laboratory results within 2 weeks prior to radiotherapy met the following criteria: ① Neutrophil count > 1,500/ MCL Heathko-Pilot Oncology Research Fund; ② Platelet > 50,000/ MCL; ③ Total bilirubin < 1.5 times of the normal upper limit value; ④AST(SGOT)/ALT(SGPT) < 2.5 times of the normal upper limit; ⑤ Serum creatinine < 1.5 times of the normal upper limit value; ⑥ The results of coagulation function examination were within the normal range
* Women of childbearing age must have taken reliable contraceptive measures or conducted pregnancy tests (serum or urine) within 7 days before admission, and the results are negative, and are willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the trial drug. For men, they must agree to use appropriate methods of contraception or surgical sterilization during the trial period and 8 weeks after the last administration of the trial drug
* Understand and voluntarily sign written informed consent
* The investigator judged that the patient had good compliance

Exclusion Criteria:

* Malignant pleural/pericardial effusions, previous thoracic radiotherapy or chemotherapy
* Uncontrolled concurrent diseases, including but not limited to symptomatic congestive heart failure, unstable angina pectoris and myocardial infarction, uncontrolled grade III hypertension, liver insufficiency, renal insufficiency, uncontrolled diabetic blood sugar, arrhythmia, mental illness or social condition, etc.
* Pregnant or nursing women
* The patient has no history of intracranial hemorrhage or spinal cord hemorrhage
* HIV-positive patients receiving combination antiretroviral therapy
* Active tuberculosis
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Prior allogeneic stem cell or solid organ transplantation
* Researchers determine other conditions that may affect the conduct of clinical studies and the determination of their findings

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced (Stage IIIa or IIIb) NSCLC that was histologically or cytologically inoperable.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of radiation respiratory events or esophagitis with grade 3 or higher | after radiation therapy，up to 1 year
  incidence of radiation respiratory events or esophagitis with grade 3 or higher

SECONDARY OUTCOMES:
objective response rate | through study completion，up to 12 weeks
  objective response rate
locate control rate | through study completion，up to 12 weeks
progression-free survival | through study completion，up to 12 weeks
overall survival | through study completion, an average of 2 year

IPD SHARING:
Plan to Share IPD: No